CLINICAL TRIAL: NCT01571778
Title: The Utility of Hand Hygiene Before Non-sterile Glove Use
Brief Title: Hand Hygiene Before Non-sterile Glove Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Kerri A Thom, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: HP-00051378
Record Dates: First submitted 2012-03-29; First posted 2012-04-05 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Hand Hygiene
Keywords: Hand Hygiene; Non-sterile Glove Use

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Donning Gloves without Hand Hygiene (Experimental): In this arm, healthcare workers will be assigned to don non-sterile gloves prior to patient contact WITHOUT first performing hand hygiene. Samples will be obtained from hands prior to donning gloves and from the gloves after donning to determine total aerobic colony counts and to identify important hospital pathogens
  Interventions: Behavioral: Hand Hygiene before Donning Non-sterile Gloves
- Hand Hygiene before donning Non-Sterile Gloves (No Intervention): In this arm, healthcare workers will be assigned to first perform hand hygiene before donning non-sterile gloves prior to patient contact (This is usual,expected practice). Samples will be obtained from hands prior to donning gloves and from the gloves after donning to determine total aerobic colony counts and to identify important hospital pathogens

INTERVENTIONS:
Behavioral: Hand Hygiene before Donning Non-sterile Gloves — In the "No Intervention" arm, healthcare workers will be assigned to first perform hand hygiene before donning non-sterile gloves prior to patient contact (usual practice). Samples will be obtained from hands prior to donning gloves and from the gloves after donning to determine total aerobic colony counts and to identify important hospital pathogens
  In the Experimental arm, they will be instructed to don gloves without washing their hands as described.
  Arms: Donning Gloves without Hand Hygiene

SUMMARY:
The importance of healthcare worker hand hygiene in decreasing bacterial transmission between patients is well documented. Healthcare workers may don non-sterile gloves in routine care of patients, particularly for those patients known or suspected to harbor epidemiologically important microorganisms. Governing bodies currently recommend performing hand hygiene prior to donning gloves and after glove removal. The importance of hand hygiene post glove removal is well shown, however few studies exist to show utility of hand hygiene prior to donning gloves. In fact, data suggests that glove use is an impediment to hand hygiene and may reduce compliance with hand washing. In light of this and the fact that no evidence exists that washing hands BEFORE glove use is important, the aim of the study is to asses the utility of routine hand hygiene prior to donning non-sterile gloves before a patient contact.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare worker engaging in direct patient contact on Contact Precautions (e.g. expected glove use)
* >= 18 years of age

Exclusion Criteria:

* Visibly soiled hands requiring hand washing (cannot randomize)
* Non-compliance with glove use as indicated for care of patient on Contact Precautions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Difference in Total Aerobic Colony Counts | The total time of participation from the healthcare worker will be approximately 2-3 minutes, the time needed to perform hand hygiene and don gloves (group 1) or don gloves (group 2).
  The Difference in Total Aerobic Colony Counts from hands at baseline (Group 1, prior to Hand Hygiene; Group 2, prior to donning gloves) to gloves after donning

SECONDARY OUTCOMES:
Pathogen Identification | The total time of participation from the healthcare worker will be approximately 2-3 minutes, the time needed to perform hand hygiene and don gloves (group 1) or don gloves (group 2).
  Gloves will be sampled from both groups after donning and evaluation for important hospital pathogens will be performed

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States